CLINICAL TRIAL: NCT06752733
Title: The Association Between Myocardial Stunning and Long-term Prognosis After Electrical Cardioversion in Patients with Atrial Fibrillation
Brief Title: Cardiac Stunning After Electrical Cardioversion
Acronym: AMPEA
Status: Active, not recruiting | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Roh Seung Young, Professor, Korea University Guro Hospital
Other Study IDs: 2020GR0213
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Atrial fibrillation: A group of patients with atrial fibrillation refractory to pharmacological treatment who are candidates for electrical cardioversion
  Interventions: Procedure: electrical cardioversion

INTERVENTIONS:
Procedure: electrical cardioversion — synchronized electrical shocks to restore normal sinus rhythm in patients with atrial fibrillation, performed under sedation

SUMMARY:
The goal of this observational study is to evaluate cardiac stunning and electrocardiographic parameters through transthoracic echocardiography and 24 hours ECG conducted immediately following electrical cardioversion. The main question it aims to answer is:

Do echocardiographic and electrocardiographic parameters relating to cardiac stunning predict atrial fibrillation (AF) recurrence rates after electrical cardioversion?

Participants will undergo echocardiography and a 24-hour Holter monitoring immediately after electrical cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation
* Patients with persistent or symptomatic atrial fibrillation who are candidates for electrical cardioversion
* Patients eligible for anticoagulation therapy for thromboembolism prevention before and after the procedure
* Patients who can understand and provide written informed consent

Exclusion Criteria:

* Patients under 18 years of age or over 80 years of age
* Patients who do not consent to participate in the study
* Patients with severe coronary artery stenosis
* Patients with severe hepatic dysfunction
* Patients with severe renal dysfunction
* Patients with severe valvular heart disease
* Patients with a high risk of severe bleeding
* Patients with a history of atrial fibrillation-related catheter ablation or cardiac surgery
* Patients with an expected life expectancy of less than 1 year
* Potentially pregnant individuals
* Patients deemed unsuitable for the study by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korea University College of Medicine, Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The recurrence of atrial arrhythmia | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Medicine Guro hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No